CLINICAL TRIAL: NCT04901234
Title: Adaptive RadioTherapy for Locally Advanced OroPharynx Cancer (ART-OPC) A Phase II Randomized Trial
Brief Title: Adaptive RadioTherapy for OroPharynx Cancer
Acronym: ART-OPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Austin Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ART-OPC
Record Dates: First submitted 2021-05-17; First posted 2021-05-25 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Oropharynx Cancer; Radiotherapy; Complications; Radiotherapy Side Effect; Dysphagia; MRI
Keywords: Oropharynx cancer; Radiotherapy; Adaptation; Magnetic resonance imaging
MeSH Terms: conditions — Oropharyngeal Neoplasms; Radiation Injuries; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Phase II open label randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard radiotherapy (Active Comparator): Radiotherapy as planned at baseline, with replanning allowed only if significant weight loss or change in anatomy due to unforeseen circumstances (eg that would affect dosimetry and treatment delivery of baseline treatment plan). No adaptation to shrinking tumour is allowed.
  Interventions: Radiation: Standard radiotherapy +/- chemotherapy
- Adaptive radiotherapy (Experimental): Systematic radiation treatment plan adaptation according to the shrinking tumour on mid-treatment MRI.
  Interventions: Radiation: Experimental radiotherapy +/- chemotherapy

INTERVENTIONS:
Radiation: Standard radiotherapy +/- chemotherapy — No radiotherapy adaptation unless major dosimetric deviation
  Arms: Standard radiotherapy
Radiation: Experimental radiotherapy +/- chemotherapy — Systemic MRI-based radiotherapy adaptation mid-treatment
  Arms: Adaptive radiotherapy

SUMMARY:
This is a phase II randomized trial, where patients with histologically proven squamous cell carcinoma of oropharynx that have primary tumor (T3 - T4) in place, treated with curative intent chemoradiation, will be randomized to systematic mid-treatment MRI-based radiotherapy adaptation vs. standard of care. The primary objective is to compare patient-rated dysphagia (as assessed by the MD Anderson Dysphagia Inventory composite score at 6 months post-treatment in patients undergoing routine mid-treatment MR-guided radiotherapy adaptation vs. in patients receiving the current standard of care.

DETAILED DESCRIPTION:
Background: Dysphagia was shown to be the main driver of adverse quality of life after head and neck radiotherapy. Over the 7-week radiotherapy course, patients with head and neck cancers undergo significant anatomical changes, including weight loss and tumor shrinkage (with complete response at mid-treatment in as high as 50% of patients). The current standard of care is to maintain the same radiotherapy plan for the entire treatment duration, unless major dosimetric deviations are detected. The use of MRI for treatment adaptation has the advantage of increased soft tissue contrast and is being integrated into several clinical practises with the recent development of MR-Linac technology. However, there is currently no demonstrated clinical advantage from the use of MRI for treatment adaptation in head and neck cancer.

Primary objective: To compare patient-rated dysphagia (as assessed by the MD Anderson Dysphagia Inventory composite score at 6 months post-treatment in patients undergoing routine mid-treatment MR-guided radiotherapy adaptation vs. in patients receiving the current standard of care.

Methods: This is a phase II randomized trial, where patients with histologically proven squamous cell carcinoma of oropharynx that have primary tumor (T3 - T4) in place, treated with curative intent chemoradiation, will be randomized to systematic mid-treatment MRI-based radiotherapy adaptation vs. standard of care. Patients with contra-indications to MRI will be excluded. The study will use a 2-sided, independent-sample t-test with an alpha level of 0.05 and power of 80%, with a 1:1 randomization between the 2 arms. In order to detect a 10-point improvement in the MD Anderson Dysphagia Index (MDADI) and assuming that the quality of life scores would be normally distributed with a standard deviation of 18, a total of 104 patients will be required (52 in each arm), which has been increased to 120 patients overall (60 patients in each arm) to account for a 10% dropout rate in completion of the quality of life scoring at 6 months post-treatment. An independent DSMB will review the pooled standard deviation of the interim data collected for this trial after 40 patients overall have been recruited (20 in each arm) the value of the standard deviation used to calculate the sample size required. The DSMB will inform the study team if there is potential to reduce the sample size if the standard deviation was much lower than 18 (i.e. <=15 would result in a reduction of 25% in patients required), which will potential reduce the length of the trial. Patients will be stratified by institution and recruited in blocks of 4 to ensure a balance between arms at the interim assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Ability to provide written informed consent.
* Stage T3-T4N0-3 as per AJCC 8th edition
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Biopsy proven diagnosis of squamous cell carcinoma of the oropharynx.
* Planned for curative radiotherapy +/- chemotherapy
* For females of child-bearing age, a negative pregnancy test
* Patients treated with induction chemotherapy can be included if they have residual tumor in place.

Exclusion Criteria:

* Previous irradiation of the head and neck (HNC) region, excluding superficial radiation therapy for non-melanomatous skin cancer
* Previous surgery of the HNC region (except for incisional or excisional biopsies)
* Pregnancy or breastfeeding
* Connective tissue disease
* Any medical condition that could, in the opinion of the investigator, prevent follow-up after radiotherapy.
* Patients with contra-indications to MRI will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient-reported dysphagia | at 6 months post treatment
  Patient-reported dysphagia as measured by the MD Anderson Dysphagia Index. Overall score ranges from 0 to 100, with higher score representing better functioning and quality of life.

SECONDARY OUTCOMES:
Acute and late toxicities | From treatment start to 5-years after the end of chemoradiation]
  Rate of grade ≥ 3 late toxicity as per CTCAE v5.0

OTHER OUTCOMES:
Locoregional control | at 6 months, 2 and 5 years
Disease-free survival | at 6 months, 2 and 5 years
Overall survival | at 6 months, 2 and 5 years
Complete response rate | at 6 months
Patient-reported dysphagia | [Time Frame: At baseline, and 1-, 3-, 12- months post-treatment, and yearly up to 5 years after the end of chemoradiation]
  Patient-reported dysphagia as measured by the MD Anderson Dysphagia Index. Overall score ranges from 0 to 100, with higher score representing better functioning and quality of life.

CONTACTS AND LOCATIONS:
Locations (2):
- Austin Health, Melbourne, Australia
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada